CLINICAL TRIAL: NCT04748900
Title: Effects of a Respiratory Physiotherapy Treatment Plan in Allergic Bronchopulmonary Aspergillosis: Case Report
Brief Title: Physiotherapy Treatment Plan in Allergic Bronchopulmonary Aspergillosis: Case Report
Status: Completed | Type: Observational
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, Principal Investigator, Universidad Católica de Ávila
Other Study IDs: 04/02/2021
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Obstructive Pulmonary Disease
Keywords: Obstructive Pulmonary Disease; Physiotherapy
MeSH Terms: conditions — Lung Diseases, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: spirometer — different values are measured on the spirometer after training in respiratory physiotherapy.

SUMMARY:
A spirometry study is performed in a patient diagnosed with allergic bronchopulmonary aspergillosis. An initial measurement is carried out and the patient is then put on a four-week physiotherapy treatment plan. Four spirometry measurements were taken to assess different variables and an improvement in all the spirometry values was established.

ELIGIBILITY:
Inclusion Criteria:

* woman
* diagnosis of respiratory insufficiency due to allergic bronchopulmonary aspergillosis
* over 50 years of age
* under 80 years of age

Exclusion Criteria:

* male
* not have a diagnosis of respiratory insufficiency due to allergic bronchopulmonary aspergillosis
* under 50 years of age
* over 80 years of age

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with respiratory insufficiency due to allergic bronchopulmonary aspergillosis
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Total volume | 3 months
  ml
Vital capacity | 3 months
  ml
Expiratory reserve volume | 3 months
  ml
Inspiratory reserve volume | 3 months
  ml
Inspiratory capacity | 3 months
  ml
Inspiration time | 3 months
  seconds
Expiratory time | 3 months
  seconds

SECONDARY OUTCOMES:
Total time | 3 months
  seconds
Percentage inspiratory time | 3 months
  seconds

CONTACTS AND LOCATIONS:
Overall Officials: Jorge V Saornil, PhD, Principal Investigator — Universidad Católica de Ávila
Locations (1):
- Universidad Católica de Ávila, Ávila, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bonaiti G, Merati V, Pesci A, Faverio P. Allergic bronchopulmonary aspergillosis screening in bronchiectasis: is there always a precise answer to a clear question? Eur Ann Allergy Clin Immunol. 2019 Jan;51(1):41-43. doi: 10.23822/EurAnnACI.1764-1489.62. No abstract available. PMID 30638358
- [Result] Cui L, Liu H, Sun L. Multidisciplinary respiratory rehabilitation in combination with non-invasive positive pressure ventilation in the treatment of elderly patients with severe chronic obstructive pulmonary disease. Pak J Med Sci. 2019 Mar-Apr;35(2):500-505. doi: 10.12669/pjms.35.2.459. PMID 31086540
- [Result] Lareau SC, Fahy B. Pulmonary Rehabilitation. Am J Respir Crit Care Med. 2018 Nov 15;198(10):P19-P20. doi: 10.1164/rccm.19810P19. No abstract available. PMID 30431331
- [Result] Patel G, Greenberger PA. Allergic bronchopulmonary aspergillosis. Allergy Asthma Proc. 2019 Nov 1;40(6):421-424. doi: 10.2500/aap.2019.40.4262. PMID 31690385
- [Result] Oguma T, Taniguchi M, Shimoda T, Kamei K, Matsuse H, Hebisawa A, Takayanagi N, Konno S, Fukunaga K, Harada K, Tanaka J, Tomomatsu K, Asano K. Allergic bronchopulmonary aspergillosis in Japan: A nationwide survey. Allergol Int. 2018 Jan;67(1):79-84. doi: 10.1016/j.alit.2017.04.011. Epub 2017 May 23. PMID 28546015
- [Result] HINSON KF, MOON AJ, PLUMMER NS. Broncho-pulmonary aspergillosis; a review and a report of eight new cases. Thorax. 1952 Dec;7(4):317-33. doi: 10.1136/thx.7.4.317. No abstract available. PMID 13015523
- [Result] Denning DW, Pleuvry A, Cole DC. Global burden of allergic bronchopulmonary aspergillosis with asthma and its complication chronic pulmonary aspergillosis in adults. Med Mycol. 2013 May;51(4):361-70. doi: 10.3109/13693786.2012.738312. Epub 2012 Dec 4. PMID 23210682
- [Result] Kalaiyarasan, Jain AK, Puri M, Tayal D, Singhal R, Sarin R. Prevalence of allergic bronchopulmonary aspergillosis in asthmatic patients: A prospective institutional study. Indian J Tuberc. 2018 Oct;65(4):285-289. doi: 10.1016/j.ijtb.2018.04.007. Epub 2018 Apr 13. PMID 30522614
- [Result] Sehgal IS, Choudhary H, Dhooria S, Aggarwal AN, Bansal S, Garg M, Behera D, Chakrabarti A, Agarwal R. Prevalence of sensitization to Aspergillus flavus in patients with allergic bronchopulmonary aspergillosis. Med Mycol. 2019 Apr 1;57(3):270-276. doi: 10.1093/mmy/myy012. PMID 29566248